CLINICAL TRIAL: NCT06826690
Title: A Comparative Factorial Study Design of Adjuvant Enhanced Ultrasound-Guided Wrist Block Anaesthesia for Hand Surgery : Bupivacane, Dexamethasone, Dexametmiodine
Brief Title: Comparative Factorial Study Design of Ultrasound Guided Wrist Block for Hand Surgery Comparing Effect of Bupivacane Alone and Bupivacane with Dexamethasone and Bupivacane with Dexametmiodine and Bupivacane with Dexamethasone and Dexametmiodine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mahmoud Rafaat Mohamed (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Rafaat Mohamed, Resident doctor, Aswan University
Organization: Aswan University (Other)
Allocation: Not Applicable | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 963-9-24
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-08

CONDITIONS: Hand Surgeries
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Group 1: ultrasound guided wrist block with bupivacane alone (Active Comparator): Group 1: ultrasound guided wrist block with bupivacane.025% .. 15 ml volume totally
- Group2: ultrasound guided wrist block with bupivacane.25% and 8mg dexamethasone (Active Comparator): Group 2: 40 patients receive ultrasound guided wrist block with 15 ml volume including bupivacane.25% and 8 mg dexamethasone
- Group 3: ultrasound guided wrist block with bupivacane and dexametmiodine (Active Comparator): Group 3: 40 patients receive ultrasound guided wrist block with 15 ml volume totally including bupivacane.25% and 50 mcg dexametmiodine
- Group 4: ultrasound guided wrist block with bupivacane and dexametmiodine and dexamethasone (Active Comparator): Group 4 : 40 patients receive ultrasound guided wrist block with 15 ml volume including bupivacane.25% and 8 mg dexamethasone and 50 mcg dexametmiodine

INTERVENTIONS:
Procedure: Group 1: ultrasound guided wrist block with bupivacane alone — Ultrasound guided wrist block with 15 ml volume of bupivacane.25%
Procedure: Group 2 : ultrasound guided wrist block with bupivacane and dexamethasone — Group 2 : patients receive ultrasound guided wrist block with bupivacane.25% and 8 mg dexamethasone.. 15 ml volume totally
Procedure: Group 3: ultrasound guided wrist block with bupivacane and dexametmiodine — Group 3 will receive ultrasound guided wrist block with bupivacane.25% and 50 mcg dexametmiodine... 15 ml volume totally
Procedure: Group 4: patients will receive ultrasound guided wrist block with bupivacane and dexamethasone and dexametmiodine — Group 4 patients will receive ultrasound guided wrist block with bupivacan.25%e and 8 mg dexamethasone and 50 mcg dexametmiodine

SUMMARY:
Ultrasound guided wrist block comparing effect of bupivacane alone and bupivacane with dexamethasone and bupivacane with dexametmiodine and bupivacane with dexamethasone and dexametmiodine

DETAILED DESCRIPTION:
Ultrasound guided wrist block comparing effect of bupivacane alone and bupivacane with dexamethasone and bupivacane with dexametmiodine and bupivacane with dexametmiodine and dexamethasone.

Taking medical and surgical history from patients. Taking base line data as heart rate and blood pressure and spo2. Measure duration of analgesia for post operative pain using NRS for 24 hours abd recording NRS at time interval of 2 , 4,6,12,24 hours post operative.

Any patient the NRS above 4 will receive 5 mg nalbufin . Recording patients satisfaction by a survey .

ELIGIBILITY:
Inclusion Criteria:

- Patients more than or equal 18 years old and are ASA 1-3

Exclusion Criteria:

* allergy to used medication
* pre exist neuropathy
* coagulapthy
* cognitive impairment
* refusal to participate
* Failed block and requiring general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-08-07 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Comparing the effectiveness of bupivacane alone and bupivacane with dexamethasone and bupivacane with dexametmiodine and bupivacane with dexamethasone and dexametmiodine | 24 hour
  Comparing duration of analgesia by each combination from block administration to first request of analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Zaher Zaki Zaher, Specialist, Study Director
Locations (1):
- Aswan university hospital, Aswān, Aswan Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided